CLINICAL TRIAL: NCT03698344
Title: Sympathetic Nerve Response Incited by Biodiesel Exhaust Exposure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Umeå University (Other)
Responsible Party: Principal Investigator, Jenny Bosson, Principal Investigator, Umeå University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Umu-2018-348-32M
Record Dates: First submitted 2018-10-04; First posted 2018-10-09 (Actual); Last update posted 2019-09-30 (Actual); Status verified 2019-09

CONDITIONS: Healthy; Exposure to Pollution
Keywords: air pollution; microneurography; MNSA; Biodiesel; RME

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Biodiesel exhaust exposure (Experimental): A single arm study in which first a filtered air baseline muscle sympathetic nerve activity (MSNA) is recorded with and without an exposure mask. When measurements have been secured exposure to dilute biodiesel exhaust will start.
  Interventions: Other: Biodiesel exhaust exposure

INTERVENTIONS:
Other: Biodiesel exhaust exposure — Evaluation of sympathetic nervous system activity as assessed by microneurography recording during an acute exposure to dilute biodiesel exhaust via mask.

SUMMARY:
The adverse effects of current ambient air pollution on cardiovascular and respiratory health have been demonstrated in an extensive series of epidemiological, observational and experimental studies. Similar cardiovascular responses seen post diesel exposure have been shown to occur following biodiesel exhaust exposure as well. In the current project the investigators aim to determine whether an acute exposure to biodiesel exhaust (rapeseed methyl ester) causes impacts on sympathetic nervous system activation in healthy volunteers.

DETAILED DESCRIPTION:
Brief as well as chronic exposures to ambient air pollution have been linked with increases in cardiovascular morbidity and mortality. Evidence suggests that the strongest associations between air pollution exposure and adverse cardiovascular effects are found for combustion-derived particulate matter, especially in the fine and ultrafine ranges such as is found in diesel engine emissions as well as biodiesel exhaust (RME, rapeseed methyl ester). Despite a greater understanding of the cardiovascular effects of air pollution, the underlying mechanism through which exposure to fine and ultrafine particulate air pollution alters vascular function has yet to be determined. Microneurography is a method that records nerve impulse traffic in human peripheral nerves, allowing for the assessment of sympathetic nervous activity. The current study will employed microneurography techniques to evaluate autonomic function in association with inhaled biodiesel exhaust exposure in healthy human volunteers.

ELIGIBILITY:
Criteria:

Inclusion Criteria:

Healthy (normal ECG, lung function, blood sample, clinical examination)

Exclusion Criteria:

Metabolic disease Cardiovascular disease Respiratory disease BMI ≥ 30 Use of psychoactive medication Infection within 2 weeks of the study Smokers or regular snus usage

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2018-10-29 (Actual); Primary Completion 2018-12-21 (Actual); Study Completion 2019-02-15 (Actual)

PRIMARY OUTCOMES:
Microneurography | 1 hour
  Microneurography recording of muscle sympathetic nervous system activity

CONTACTS AND LOCATIONS:
Overall Officials: Jenny A Bosson, MD;PhD, Principal Investigator — Umeå University
Locations (1):
- Dept of Medicine, Lung and Allergy section, University Hospital, Umeå, Sweden

IPD SHARING:
Plan to Share IPD: Undecided